CLINICAL TRIAL: NCT01429805
Title: Balloon Assisted Hip Arthroscopy - Clinical Evaluation of a New Tool for Hip Arthroscopy
Acronym: BAHA-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pivot Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PR01662
Record Dates: First submitted 2011-09-05; First posted 2011-09-07 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Hip Arthroscopy
Keywords: Hip arthroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: HipJack Balloon Spacer — Use of the HipJack Kit to maintain distraction of the joint during hip arthroscopy.

SUMMARY:
The purpose of this study is to obtain information on the safety and performance of HipJack Balloon Spacer to access the central compartment of the hip and maintain intra-articular hip joint distraction during arthroscopy of the central compartment of the hip.

DETAILED DESCRIPTION:
The HipJack Kit is intended to maintain distraction of the joint during hip arthroscopy. This study will evaluate the Kit in clinical sites outside of the United States.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled for unilateral arthroscopic procedure of the hip

Exclusion Criteria:

* Active infection sepsis or osteomyelitis
* Body mass index (BMI) of 40 or greater
* Open wounds of the hip or leg area
* Moderate or severe degenerative hip disease or hip joint space <3 mm
* Large pincer, coxa profunda or protrusio
* Retroverted acetabulum
* Compromised ligamentum teres or ligamentum teres dysplasia
* Previous hip surgery or arthroscopy on the target hip
* Hip injury due to high-energy trauma
* Hip fracture or hip dislocation on the target hip
* Metabolic disorders that may impair bone formation
* Osteomalacia or moderate to severe osteoporosis, rapid joint destruction, marked bone loss or bone resorption noted on x-ray
* Severe neurosensory deficits
* Inadequate joint space distraction with external traction to allow for insertion of HipJack device
* Any condition that is a relative or absolute contraindication to hip arthroscopy
* Pregnant or lactating
* History of venous thrombosis or known coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Ability to access the central compartment of the hip and maintain intra-articular hip joint distraction with the HipJack Balloon Spacer during hip arthroscopy. | Treatment (Day 0)

SECONDARY OUTCOMES:
Reduction in external traction time. | Treatment (Day 0)
Investigator-related adequacy of central compartment visualization with use of the investigational device. | Treatment (Day 0)
Investigator-rated adequacy of maneuverability of arthroscopy tools with the investigational device inflated in the central compartment. | Treatment (Day 0)
The occurrence of serious adverse events by 6-week follow-up rated by the investigator to be probably or definitely related to the investigational device. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Ramachandran, MD, Principal Investigator — Barts and The London NHS Trust
Locations (3):
- UZ Leuven, Pellenberg, Belgium
- Schulthess Clinic, Zurich, Switzerland
- Barts and The London NHS Trust, London, United Kingdom